CLINICAL TRIAL: NCT00880373
Title: An Evaluation of the Effectiveness of Ibuprofen and Opioid (Morphine or Diamorphine) for Acute Pain in Sickle Cell Disease: a Double-blind, Placebo-controlled Randomised Trial
Brief Title: Ibuprofen and Opioid (Morphine or Diamorphine) for Acute Pain in Sickle Cell Disease - Sickle With Ibuprofen & Morphine
Acronym: SWIM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The funding withdrawal and early termination of the trial is based upon lack of suitable recruitment figures in order to reach the required trial endpoints.
Sponsor: London North West Healthcare NHS Trust (Other)
Collaborators: Medical Research Council CTU (Unknown)
Responsible Party: Dr Kofi Anie, North West London Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTA 07/48/01; ISRCTN97241637
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Pain; Ibuprofen; Morphine; Diamorphine; Patient Controlled Analgesia
MeSH Terms: conditions — Anemia, Sickle Cell; Pain | interventions — Ibuprofen; Heroin; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Diamorphine or Morphine by PCA and oral ibuprofen
  Interventions: Drug: Ibuprofen; Drug: Diamorphine or Morphine
- 2 (Placebo Comparator): Diamorphine or Morphine by PCA and oral placebo
  Interventions: Drug: Placebo; Drug: Diamorphine or Morphine

INTERVENTIONS:
Drug: Ibuprofen — Oral ibuprofen 800 mg three times daily for a total of 2400 mg per day for 4 days
  Arms: 1
Drug: Placebo — Matching placebo three times daily for 4 days
  Arms: 2
Drug: Diamorphine or Morphine — Diamorphine or Morphine by PCA

SUMMARY:
The use of oral ibuprofen combined with Opioid (Morphine or Diamorphine) administered through patient controlled analgesia (PCA) will be clinically effective for acute pain crisis in adults with sickle cell disease (SCD).

DETAILED DESCRIPTION:
Pain from vaso-occlusion in sickle cell disease (SCD) is persistent, and its management continues to pose a challenge to practitioners. Opioids are recommended for the treatment of severe acute SCD pain, and have been used successfully within the hospital setting. Non-steroidal Anti-Inflammatory Drugs (NSAIDs) are recommended for acute SCD pain, however there is no clear evidence for the effectiveness of oral NSAIDs in combination with parenteral opioids in adults with SCD.Data from acute pain research suggests that oral ibuprofen is one of the best NSAIDs for combination treatment with morphine via PCA.

This is a randomised controlled trail to evaluate the effectiveness of oral ibuprofen plus intravenous Diamorphine or morphine via PCA. The results will provide the evidence needed to recommend whether or not ibuprofen should be used in acute SCD pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with SCD of any phenotype

Exclusion Criteria:

* Patient has a history of allergic reaction to either diamorphine/morphine or ibuprofen
* Patient has contraindications to diamorphine/morphine or ibuprofen, e.g. peptic ulcer disease, non-steroidal anti-inflammatory drug (NSAID)-induced asthma
* Patient in a drug dependency programme
* Patient is on renal dialysis
* Stroke within the last 6 weeks
* Platelet count less than 50 x 10^9/l
* Patient is pregnant or breastfeeding
* Doctor unwilling to randomise the patient for other reasons
* Previous participation in the trial
* Patient receiving drug treatment with which opioids or NSAIDs are likely to interact significantly
* Stage 1 - 5 chronic kidney disease (ref Appendix 2), including urine protein: creatinine ratio of >50 (Because the ibuprofen dose is substantial it is felt that precautions should be taken to exclude those who have any signs of chronic kidney disease. One of the signs of kidney disease is "persistent proteinuria". Therefore, the patient who intermittently has proteinuria(which could be due to other reasons) could still participate.)
* Oxygen saturation by pulse oximetry <94%
* Participation in another clinical trial within the last month

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Patient controlled analgesia (PCA)diamorphine or morphine consumption | 4 days

SECONDARY OUTCOMES:
Rapidity of pain control - time to achieve a pain score of 4 on a standard 10-point numeric rating scale | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Kofi A Anie, PhD, Principal Investigator — London North West Healthcare NHS Trust; Gavin Cho, MD, Study Chair — London North West Healthcare NHS Trust; Mark Layton, MD, Principal Investigator — Imperial College London; Sarah Meredith, MD, Study Director — MRC Clinical Trials Unit; Caroline Dore, BSc, Study Director — MRC Clinical Trials Unit
Locations (2):
- United Kingdom (2):
  - North West London Hospitals NHS Trust, London
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Derived] Cho G, Anie KA, Buckton J, Kiilu P, Layton M, Alexander L, Hemmaway C, Sutton D, Amos C, Dore CJ, Kahan B, Meredith S. SWIM (sickle with ibuprofen and morphine) randomised controlled trial fails to recruit: lessons learnt. BMJ Open. 2016 Jun 9;6(6):e011276. doi: 10.1136/bmjopen-2016-011276. PMID 27288381